CLINICAL TRIAL: NCT06260683
Title: A Comprehensive Evaluation of Tobacco-Flavored vs. Non-Tobacco Flavored E-Cigarettes on Smoking Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Theodore Wagener, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-22240; NCI-2023-04102 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01DA057327 (NIH)
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Arm I (PEC) (Experimental): Participants receive PEC for 14 weeks, including a 2-week pre-switch period to become familiar with usage. Participants in all arms participate in discussions throughout the trial.
  Interventions: Other: Questionnaire Administration; Device: Vaping
- Arm II (TEC) (Experimental): Participants receive TEC for 14 weeks, including a 2-week pre-switch period to become familiar with usage. Participants in all arms participate in discussions throughout the trial.
  Interventions: Other: Questionnaire Administration; Device: Vaping
- Arm III (NRT) (Active Comparator): Participants receive NRT (nicotine patches and lozenges) for 14 weeks, including a 2-week pre-switch period to become familiar with usage. Participants in all arms participate in discussions throughout the trial.
  Interventions: Drug: Nicotine Replacement; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Nicotine Replacement — Given nicotine patches and nicotine lozenges
  Other Names: Nicotine Replacement Therapy; NRT
  Arms: Arm III (NRT)
Other: Questionnaire Administration — Ancillary studies
Device: Vaping — Given Preferred Flavor e-liquid
  Other Names: Vape
  Arms: Arm I (PEC)
Device: Vaping — Given Tobacco flavored e-liquid
  Other Names: Vape
  Arms: Arm II (TEC)

SUMMARY:
This clinical trial compares the use of tobacco flavored electronic cigarettes (ECs) vs. non-tobacco flavored ECs vs. nicotine replacement therapy (patches and lozenges) on smoking behavior in current cigarette smokers. ECs may reduce cigarette craving and withdrawal symptoms, increase motivation and confidence to stop cigarette smoking, and decrease cigarette smoking and dependence. By comparing participants' preferred flavor ECs (PEC) to tobacco flavor ECs (TEC) to NRT, researchers hope to determine the effect of EC flavors on appeal and use and learn how ECs affect smoking behaviors and health.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine PEC versus vs. TEC vs. nicotine replacement therapy (NRT) on tobacco use patterns including product switching, abstinence from cigarettes, and number of cigarettes smoked.

II. Examine PEC vs. TEC vs. NRT on cigarette craving, withdrawal symptoms, and perceived nicotine dependence.

III. Examine PEC vs. TEC on product appeal and uptake, including initial trial, days used during period of product provision, and purchase and continued use after 12 weeks.

OUTLINE: Participants are randomized to 1 of 3 arms.

ARM I: Participants receive PEC for 14 weeks, including a 2-week pre-switch period to become familiar with usage.

ARM II: Participants receive TEC for 14 weeks, including a 2-week pre-switch period to become familiar with usage.

ARM III: Participants receive NRT (nicotine patches and lozenges) for 14 weeks, including a 2-week pre-switch period to become familiar with usage.

Participants in all arms participate in discussions throughout the trial.

SURVEILLANCE PHASE: Participants in all arms are followed for 12-weeks after completion of study procedures.

ELIGIBILITY:
Inclusion Criteria:

* >= 21 years old
* Smoke >= 5 cigarettes per day for the past year
* Willing to use either an EC or NRT
* Read and speak English
* Have a smartphone

Exclusion Criteria:

* Report currently using smoking cessation medications, NRT, or actively seeking treatment for smoking cessation
* Current use of an EC > 4 days a month
* Diagnosed medical conditions of lung disease, asthma, cystic fibrosis, heart disease or chronic obstructive pulmonary disease (COPD)
* Unmanaged (unmedicated and/or without counseling) diagnosis of schizophrenia
* History of cardiac event or distress within the past 3 months
* Currently pregnant, planning to become pregnant within 6 months, or breastfeeding
* High blood pressure not controlled by medications
* Serious angina pectoris or chest pain
* Stroke within the past three months
* Known allergy to propylene glycol or vegetable glycerin
* Serious underlying arrhythmias, irregular heartbeat or abnormal heart rhythm
* Live in same household as another study participant

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2028-04-12 (Estimated); Study Completion 2028-04-12 (Estimated)

PRIMARY OUTCOMES:
7-day point prevalence complete switching rate | At week 14
  Self-reported 7-day point prevalence abstinence (no cigarettes, not even a puff, in the previous 7 days), any reported use of ECs or NRT over the past 7 days, and an exhaled CO reading of ≤6ppm.
Biochemically verified 7-day point prevalence abstinence from cigarettes | At week 14
  Biochemical verification of abstinence from cigarettes (exhaled CO reading of ≤6ppm) combined with self-reported 7-day point prevalence abstinence (no cigarettes, not even a puff, in the previous 7 days).
Cigarettes smoked per day | At week 14
  Cigarettes smoked per day as evaluated with the timeline follow-back questionnaire.

SECONDARY OUTCOMES:
Change in cigarettes smoked per day | From baseline to 26 weeks
  Changes in cigarettes smoked per day from baseline to 26 weeks will be evaluated with the timeline follow-back questionnaire.
Change in nicotine dependence | From baseline to 14 weeks
  Among participants abstaining from smoking, changes in nicotine dependence from baseline to 14 weeks will be assessed in the PEC, TEC, and NRT arms with the PROMIS nicotine dependence scale. Scores range from 0 to 16 with higher scores indicating greater dependence.
Changes in cigarette craving and nicotine withdrawal | At baseline, 2, 6, 14, and 26 weeks
  Cigarette craving and nicotine withdrawal will be measured using the Mood and Physical Symptoms Scale (MPSS). Total MPSS scores range from 12 to 60 with higher scores indicating a greater severity of tobacco withdrawal symptoms.
Number of days used in past week | At 2, 6, and 14 weeks
  The number of days the study products are used in the past 7 days during the period of product provision in the PEC and TEC arms.
Number of days used in past month | At 6 and 14 weeks
  The number of days the study products are used in the past 30 days during the period of product provision in the PEC and TEC arms.
Product appeal | At 2, 6, 14, and 26 weeks
  EC appeal is measured with the modified Cigarette Evaluation Questionnaire (mCEQ) to assess subjected responses to ECs (e.g., reward, satisfaction).
Continued use of ECs | From 14 to 26 weeks
  The proportion of participants who continue to use ECs between 14 and 26 weeks in the PEC and TEC arms.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore L Wagener, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu